CLINICAL TRIAL: NCT04754334
Title: A Double-Blind, Placebo-controlled, Multi-center Randomized, Phase 3 Study to Evaluate the Efficacy and Safety of ORMD-0801 in T2DM Subjects With Inadequate Glycemic Control on Diet Control Only or on Diet Control and Metformin Monotherapy.
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of ORMD-0801 in Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The ORA-D-013-2 protocol was terminated based on the primary results analyzed at week 26 in the ORA-D-013-1 protocol.
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-013-2
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ORMD-0801; Insulin; Fish Oils

STUDY DESIGN:
Intervention Model Description: Approximately 450 US- and Europe-based adult male and female subjects with T2DM will be randomized in a 1:1 ratio to receive either ORMD-0801 8 mg QD (one 8 mg capsule, dosed at night), or placebo dosed QD (dosed at night). It is anticipated that 225 subjects will be randomized to each arm of the study to complete approximately 200 subjects in each arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Approximately 450 US- and Europe-based adult male and female subjects with T2DM will be randomized in a 1:1 ratio to receive either ORMD-0801 8 mg QD (one 8 mg capsule, dosed at night), or placebo dosed QD (dosed at night). It is anticipated that 225 subjects will be randomized to each arm of the study to complete approximately 200 subjects in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo dosed QD
  Interventions: Other: Placebo
- ORMD-0801 (Experimental): ORMD-0801 8 mg QD
  Interventions: Drug: ORMD-0801

INTERVENTIONS:
Drug: ORMD-0801 — Oral Insulin
  Other Names: Oral Insulin
  Arms: ORMD-0801
Other: Placebo — Fish Oil
  Other Names: Fish Oil
  Arms: Placebo

SUMMARY:
This double-masked placebo-controlled study will include approximately 450 subjects with inadequately controlled T2DM on diet control alone or on diet control and metformin monotherapy. Subjects will undergo an initial 21-day Screening Period, followed by a 26-week Double-Blind Treatment Period and a Double-Blind 26-week Treatment Extension Period.

DETAILED DESCRIPTION:
Screening Period The investigator will review the aim of the study, study procedures, potential risks, and benefits with the volunteers. These subjects will then sign a written informed consent during Screening Visit 1. They will be instructed to return to the clinic 10 days prior to randomization (Visit 1) for Screening Visit 2. At this visit, a continuous glucose monitoring (CGM) sensor will be placed with appropriate instructions by the study team for a 10-day blinded CGM data collection by the site. Subjects will then return to the clinic after 10 days (± 1-day) for removal of the CGM sensor. The subjects will be randomized to one of the three study treatment arms.

26-Week Double-Masked Treatment Period After the Screening Period, subjects will be randomized to 26 weeks of the Double-Blind Treatment Period consisting of ORMD-0801 8 mg (1 x 8 mg capsule), or placebo in a 1:1 randomized fashion. Medication will be administered once daily at night prior to bedtime (between 8 PM to 12 Midnight and no sooner than 1 hour after dinner).

During the Double-Masked Treatment Period commencing at Week 0 (Visit 1, CGM removal), subjects will return to the clinic at the following intervals: Week 6 - Visit 2; Week 12 -Visit 3; Week 18 - Visit 4; Week 24 - Visit 5 (10 days prior to Week 26 for CGM application) and Week 26 - Visit 6 (CGM removal and end of Double-Blind Treatment Period visit).

The visit requiring CGM application will occur 10 days prior to the CGM removal visit within a ± 1-day window

26-Week Double-Masked Treatment Extension Period Following the completion of the Double-Blind Treatment Period, subjects will enter a 26-week Double-Blind Treatment Extension Period. Subjects will remain on the same treatment regimen and continue to receive the same medication for the duration of the Double-Blind Treatment Extension Period. The Extension Period treatment assignments will remain blinded for the duration of the study.

Visits will occur at the following intervals during the 26-Week Double-Masked Treatment Extension Period: Week 30 - (Visit 7); Week 40 - Visit 8; Week 50 - Visit 9 (10 days prior to Week 52 for CGM application); and Week 52 - Visit 10 (CGM removal and end of Double-Blind Treatment Extension Period visit).

The visit requiring CGM application will occur 10 days prior to the CGM removal visit within a ± 1-day window.

All subjects completing the trial will return to the clinic in 2 weeks ± 3 days for a Safety Follow-Up Visit. Subjects withdrawing prematurely from the trial, will have the early termination (ET) visit procedures completed. All patients will continue to be followed in accordance with ITT principles to avoid a loss to follow-up and missing data.

ELIGIBILITY:
Inclusion Criteria:

* 1. Established diagnosis of T2DM for at least 6 months prior to Screening AND an A1C ≥ 7.5% but ≤ 11.0% at Screening.
* 2. Subjects should be on:

  * a. Diet and exercise therapy with no oral or injectable glucose lowering therapy for a period of at least 3 months prior to screening; OR
  * b. Diet and exercise therapy with a stable dose of metformin only (≥1500 mg or maximal tolerated dose) for a period of at least 3 months prior to Screening.
* 3. Body mass index (BMI) of 25-40 kg/m2 at Screening and stable weight, with no more than 5 kg gain or loss in the 3 months prior to Screening.
* 4. Renal function - GFR ≥ 30 ml/min/1.73 m2.
* 5. Females of childbearing potential must:

  * a. have a negative serum pregnancy test result at Screening.
  * b. agree to avoid becoming pregnant while receiving IP for at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP.
  * c. agree to use an acceptable method of contraception at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP. Acceptable methods of contraception are hormonal contraception (contraceptive pill or injection) PLUS an additional barrier method of contraception such as a diaphragm, condom, sponge, or spermicide.
  * d. In the absence of hormonal contraception, double-barrier methods must be used which include a combination of any two of the following: diaphragm, condom, copper intrauterine device, sponge, or spermicide, and must be used for at least 30 days prior to administration of IP, during the entire study, and for 30 days following their last dose of IP.
  * e. Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ERCs/IRBs. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.
  * f. Females who are not of childbearing potential are defined as:

    * i. Postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age); OR
    * ii. Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; OR
    * iii. Have a congenital or acquired condition that prevents childbearing.

Exclusion Criteria:

* Subjects with:
* 1. Type 1 diabetes.
* 2. A history of diabetes mellitus with ketoacidosis or is assessed by the Investigator as possibly having type 1 diabetes mellitus confirmed by a C-peptide < 0.4 ng/mL (0.13 nmol/L) at Screening.
* 3. Diabetes attributable to other secondary causes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
* 4. Concomitant treatment involving insulin, and any other inhaled, oral or injectable antihyperglycemic agents including alpha glucosidase inhibitor, meglitinides, sulfonylurea, DPP-4 inhibitor, SGLT-2 inhibitor, thiazolidinedione or GLP-1 agonists, and pramlintide within 2 months prior to Visit 1.
* 5. A history of >2 episodes of severe hypoglycemia within 6 months prior to Screening.
* 6. A history of hypoglycemic unawareness.
* 7. A history of unstable angina or myocardial infarction within 6 months prior to Screening, New York Heart Association (NYHA) Grade 3 or 4 congestive heart failure (CHF), valvular heart disease, ventricular cardiac arrhythmia requiring treatment, pulmonary hypertension, cardiac surgery, coronary angioplasty, stroke or transient ischemic attack (TIA) within 6 months prior to Screening.
* 8. A history of uncontrolled or untreated severe hypertension defined as systolic blood pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 100 mmHg. A single repeat measurement will be permitted.
* 9. Renal dysfunction: GFR < 30 mL/min/1.73 m2.
* 10. Active proliferative retinopathy requiring treatment.
* 11. Psychiatric disorders that, per Investigator judgment, may have impact on the safety of the subject or interfere with subject's participation or compliance in the study.
* 12. Laboratory abnormalities at Screening including:

  * a. C-peptide < 0.4 ng/mL.
  * b. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or >1.5X the upper limit of normal; a single repeat test is allowable.
  * c. Elevated liver enzymes (alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP)) >3X the upper limit of normal; a single repeat test is allowable.
  * d. Very high fasting triglyceride levels (>600 mg/dL); a single repeat test is allowable.
  * e. Any relevant abnormality that would interfere with the efficacy or the safety assessments during study treatment administration.
* 13. Positive history of active liver disease (other than non-alcoholic hepatic steatosis), primary biliary cirrhosis, or active symptomatic gallbladder disease.
* 14. Positive results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus ribonucleic acid (RNA).
* 15. Patient has active or history of neoplastic disease (except for adequately treated non-invasive basal cell and/or squamous cell carcinoma or carcinoma in situ of the cervix) within the past 5 years prior to Baseline.
* 16. Use of the following medications:

  * a. History of use of any injectable or inhaled, basal, pre-mixed or prandial insulin (greater than 7 days) within 6 months prior to Screening.
  * b. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening.
  * c. Requirements (in the last 12 months), or may require, systemic (oral, intravenous, intramuscular) glucocorticoid therapy for more than 2 weeks during the study period. Intra-articular and/or topical corticosteroids are not considered systemic.
  * d. Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and immunosuppressive or immunomodulating agents. Inhaled nasal steroids are permissible.
* 17. Known allergy to soy.
* 18. Involvement in a weight loss program and is not in the maintenance phase, or subject has started weight loss medication (e.g., orlistat or liraglutide) within 3 months prior to Screening.
* 19. Prior bariatric surgery.
* 20. Subject is pregnant or breast-feeding.
* 21. Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy Oramed Ltd. Protocol No. ORA-D-013-2 Phase 3 Clinical Study October 12, 2020 Page 12 alcohol intake as defined by >3 drinks per day or >14 drinks per week or binge drinking) at Screening. Occasional intermittent use of cannabinoid products will be allowed provided that no cannabinoid products have been used during the 1 week prior to each visit.
* 22. Contraindications to metformin use as per label.
* 23. A history of gastrointestinal disorders (e.g. hypochlorhydria) with the potential to interfere with drug absorption.
* 24. Any condition or other factor (at the Investigator's discretion) that is deemed unsuitable for subject enrollment into the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Mean change in A1C | Baseline and Week 26
  mean change from baseline (Visit 1) in A1C at 26 weeks (Visit 6) for the active and placebo groups. Randomization will occur at Visit 1 (Week 0),

SECONDARY OUTCOMES:
The mean change in fasting plasma glucose | baseline and week 26
  The mean change from baseline (Visit 1) in fasting plasma glucose at 26 weeks (Visit 6)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kidron, PhD, Study Chair — Oramed, Ltd.
Locations (1):
- Research Institute of South Florida, Inc. (PHARMASEEK), Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No